CLINICAL TRIAL: NCT06223503
Title: Reducing Chronic Opioid Use Among Veterans Undergoing Community Care Surgery Using a Transitional Pain Service
Brief Title: VA Transitional Pain Service Study
Acronym: VATPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 22-062
Record Dates: First submitted 2024-01-11; First posted 2024-01-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Opioid Use
Keywords: Post-operative pain; Opioid use disorder; Opioid misuse; MISSION Act; Community Care; Transitional Care Coordination
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Veterans will be randomized to either be enrolled into the Salt Lake City VAMC transitional pain service or to receive only the usual care through the community care surgeon.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth Transitional Pain Service + Standard Postoperative Follow-Up Care (Experimental): Telehealth Transitional Pain Service + Standard Postoperative Follow-Up Care
  Interventions: Behavioral: Transitional Pain Service
- Standard Follow Up Care (Active Comparator): Standard Follow Up Care
  Interventions: Behavioral: Transitional Pain Service

INTERVENTIONS:
Behavioral: Transitional Pain Service — The Transitional Pain Service (TPS) is a novel perioperative surgical home approach that consists of comprehensive pain management and care coordination before, during and for at least 6-months after surgery for Veterans at risk for chronic opioid use (COU).

SUMMARY:
The VA Community Care Program has provided an important resource to improve access to surgical care for Veterans unable to have treatment at VA Medical Centers (VAMC). However, there is an increased risk of developing chronic opioid use when at-risk surgical patients receive opioids from non-VA providers. A multidisciplinary approach to perioperative pain management known as the Transitional Pain Service (TPS) has been shown to effectively reduce chronic opioid use among Veterans after surgery, but it is unknown whether it can be used to achieve the same outcomes for Veterans using Community Care for high-risk surgery. Through this project, the investigators will generate important data to establish whether a telehealth TPS approach can serve as a scalable and effective strategy to ensure safe opioid use among Veterans undergoing orthopedic surgery. The investigators will randomize Veterans using Community Care for orthopedic surgery to telehealth TPS versus standard of care. Finally, the investigators will interview patients using Community Care to better understand barriers and facilitators to telehealth TPS and Veteran satisfaction with the approach to pain management.

DETAILED DESCRIPTION:
The Transitional Pain Service (TPS) is a novel perioperative surgical home approach that consists of comprehensive nurse care coordination before, during and for at least 6-months after surgery for Veterans at risk for chronic opioid use (COU). This program is specifically focused on 1) reducing suffering from pain and improving functional recovery after surgery; 2) preventing the development of new COU after surgery; and 3) assisting patients already on chronic opioids to taper and completely transition off narcotics during their recovery from surgery. Veterans on chronic opioids, or those identified to be at risk for persistent opioid use after surgery, are enrolled into TPS where a personalized pain management plan is developed and followed until opioid tapering is complete, or until a warm handoff can be made to their VA Primary Care Provider (PCP) to ensure continuity of care. Each Veteran's individualized pain management plan can be viewed on a SharePoint health information technology dashboard that provides clinical decision support to all VA health care providers (i.e., TPS nurse care coordinators, surgeons, VA PCPs, etc.) who provide care before and after surgery (Figure 1). Pain management and opioid use for all patients enrolled into TPS is assessed at baseline and after surgery using morphine equivalent daily dose (MEDD), and patient-reported outcomes using measures from the Patient-Reported Outcome Measurement System (PROMIS) for pain intensity (PROMIS 3a), pain interference (PROMIS 6b), and a pain catastrophizing scale (PCS) score. The TPS approach utilizes numerous evidence-based strategies that can be applied during the preoperative and postoperative period as a means to reduce opioid use and prevent CPSP among Veterans undergoing surgery at non-VA community hospitals. This includes individually tailored programs for preoperative education or pain management planning; referral for non-pharmacologic modalities such as cognitive based intervention; as well as a coordinated approach to post-discharge instructions and transitions of care. Each of these individual strategies by themselves has been shown to have an effect on improving postoperative pain management, and each is supported by current professional guidelines for the management of postoperative pain.

For Aim 1, the investigators will use claims data for opioid prescriptions submitted by non-VA surgeons across nationwide hospitals captured using the Program Integrity Tools (PIT) system for Office of Community Care data (2018-2020), and compare to pharmacy claims data for opioids prescribed to Veterans who underwent orthopedic surgery at VAMC. A risk-adjusted analysis will help determine whether non-VA surgeons are prescribing a higher quantity of opioids after surgery than VA providers. For Aim 2, the investigators will randomize Veterans from two VA medical centers who are referred for orthopedic surgery using Community Care to a transitional pain service with regular follow-up telehealth visits after surgery versus standard care. For Aim 3, the investigators will perform a qualitative study to determine what components of the telehealth TPS intervention have the greatest impact on reducing opioid use and increasing tapering after surgery at non-VA hospitals, and how often are these interventions being used as part of standard post-operative care? Semi-structured interviews will be conducted among Veterans who underwent orthopedic joint surgery at non-VA hospitals, both with and without the telehealth TPS intervention, to examined post-operative opioid usage and identify specific factors that facilitated or impeded opioid tapering.

ELIGIBILITY:
Inclusion Criteria:

Aims 1 & 3:

* The investigators will include Veterans who are referred to the Veteran Community Care Program (VCCP) for an orthopedic surgery procedure from any VA medical center throughout VISN-19.
* Additionally, these Veterans must be 18+ years of age who are not on chronic opioids at the time of surgery, and who have a VA primary care provider (PCP).

Aim 2:

* Veterans who received TPS (Aim 1) and referring VA Primary Care Providers.

Exclusion Criteria:

Aim 1:

* The investigators will exclude Veterans who are scheduled for other types of surgical procedures, are on chronic opioid therapy before surgery, are on hospice or end-of-life care, are cognitively impaired, or unable to complete the follow-up visits for any other reason.

Aim 2:

* The investigators will exclude Veterans not randomized to the TPS Telehealth intervention of Aim 1.

  * Primary Care Providers will be excluded if they do not primarily work at the VA.

Aim 3:

* The investigators will exclude Veterans who were not randomized to the TPS Telehealth intervention.
* Veterans who experienced a major complication during the perioperative period or experienced an extended length of stay (LOS) based on exceeding the upper interquartile range of median LOS.
* Exclusion criteria for this aim also include patients on hospice care, individuals discharged to a care facility, and those with scheduled readmissions for follow up procedure(s) within 90-days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Persistent post-surgical opioid use | 90 days after surgery
  The percentage of non-chronic opioid use Veterans who continue post-surgical use past 90 days after surgery.

SECONDARY OUTCOMES:
Quantity of opioids prescribed (MME/day) | 90 days after surgery
  Number of opioid tablets prescribed at discharge and in the first 90-days after surgery.
PROMIS Assessment of Pain Intensity and Pain Interference | 7, 30, 60, and 90-days after surgery
  Pain and functional patient reported outcomes using the NIH PROMIS Assessment of Pain Intensity (3a) and Pain Interference (6b). Reported as T-scores, where the average is a score of 50 and standard deviations are 10 points. A higher score represents worse pain/pain interference.
Assessment of Care Coordination | 7 days after surgery
  Assessment of care coordination during transitions using the Care Transitions Measure (CTM-15). All questions use a five-point Likert response scale comprising 'strongly disagree', 'disagree', 'neutral', 'agree' and 'strongly agree'. A single total score ranging from 0 to 100 is calculated from the CTM-15, with higher scores indicating better care transition.
Visit with Primary Care Provider within 30 days after surgery. | 30 days after surgery
  Determination of whether Veterans had a visit with their Primary Care Provider within 30 days after surgery. This is a yes/no outcome.
Number of opioid refills after discharge from surgery | Between discharge from surgery and 90-days after surgery
  The number of opioid prescription refills received after discharge from surgery and by 90-days after surgery.
Number of opioid tablets used in the 90 days after surgery | 90 days after surgery
  The difference between the number of tablets prescribed and the number of tablets left over as reported by the patient at 90 days after surgery.
Date of last opioid use | 90 days after surgery
  The date that the patient last used an opioid medication after surgery, as reported by the patient. This will be asked at days 7, 30, 60, and 90 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Brooke, MD PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yoo M, Buys MJ, Nelson RE, Patel S, Bayless KM, Anderson Z, Hales JB, Brooke BS. Effect of Multidisciplinary Transitional Pain Service on Health Care Use and Costs Following Orthopedic Surgery. Fed Pract. 2023 Dec;40(12):418-425. doi: 10.12788/fp.0438. Epub 2023 Dec 12. PMID 38812900
- [Result] Buys MJ, Anderson Z, Bayless K, Zhang C, Presson AP, Hales J, Brooke BS. Postsurgical opioid prescribing among veterans using community care for orthopedic surgery at non-VA hospitals compared to a VA hospital with a transitional pain service: a retrospective cohort study. Reg Anesth Pain Med. 2025 Jul 4;50(7):531-537. doi: 10.1136/rapm-2023-105162. PMID 38677883
- [Result] Arnaoutakis DJ, Nguyen T, Zheng X, Mao J, Patel S, Matar AH, Brooke BS, Bismuth J, Stone DH, Scali ST. Large endograft diameter is associated with poor outcomes following thoracic endovascular aortic aneurysm repair in Medicare beneficiaries. J Vasc Surg. 2025 Dec;82(6):1947-1956.e3. doi: 10.1016/j.jvs.2025.06.030. Epub 2025 Jun 26. PMID 40581193
- [Result] Brooke BS, Bayless K, Anderson Z, Holeman TA, Zhang C, Hales J, Buys MJ. Opioid tapering after surgery and its association with patient-reported outcomes and behavioral changes: a mixed-methods analysis. Reg Anesth Pain Med. 2024 Oct 8;49(10):699-707. doi: 10.1136/rapm-2023-104807. PMID 37865394